CLINICAL TRIAL: NCT04190628
Title: A Phase I, First-In-Human, Multicenter, Open-Label Dose Escalation and Dose Expansion Study of ABM-1310, as a Monotherapy and a Combination Therapy, Administered Orally in Adult Patients With Advanced Solid Tumors Harboring BRAF Mutations
Brief Title: Safety and Tolerability of ABM-1310 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Not related to safety concerns or lack of efficacy
Sponsor: ABM Therapeutics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABM1310X1101
Record Dates: First submitted 2019-12-03; First posted 2019-12-09 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumor; BRAF V600 Mutation
Keywords: Melanoma; Colorectal Cancer; Glioblastoma; Cholangiocarcinoma; Non-small Cell Lung Cancer; Thyroid Cancer; Ovarian Cancer
MeSH Terms: conditions — Melanoma; Colorectal Neoplasms; Glioblastoma; Cholangiocarcinoma; Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms; Ovarian Neoplasms | interventions — cobimetinib

STUDY DESIGN:
Intervention Model Description: Study consists of Three Parts:
  Part A: ABM-1310 Dose Escalation and MTD/RP2D Dose Confirmation
  Part B: Combination agent (ABM-1310 and cobimetinib (Cotellic®)) Dose Escalation and MTD/RP2D Dose Confirmation
  Part C: Dose Expansion (ABM-1310 Monotherapy/Combination Therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Monotherapy Dose Escalation (Experimental): A classic "3+3" design will be used to determine MTD and RP2D. Three to six patients per treatment cohort will be assigned to receive sequentially higher oral doses of ABM-1310 on a twice daily schedule (bid) for 28-day cycles, starting at a dose of 25 mg bid. Patients will receive twice daily oral doses of ABM-1310 continuously until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion is met.
  Interventions: Drug: ABM-1310
- Combination Therapy Dose Escalation (Experimental): A classic "3+3" design will guide the dose escalation in Part B. At each dose level, ABM-1310 will be administered in combination with cobimetinib (Cotellic ®) once daily (qd) for the first 21 days of each 28-day treatment cycle. The starting dose of ABM-1310 will be a dose below the MTD that has been demonstrated to be safe in Part A Monotherapy.
  Interventions: Drug: ABM-1310; Drug: Cobimetinib
- Monotherapy Therapy Dose Expansion-1 (Experimental): - In C-1(Monotherapy - Primary CNS Tumors), continuous twice daily oral doses of ABM-1310 at the recommended phase 2 dose (RP2D) from Part A until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion is met.
  Interventions: Drug: ABM-1310
- Monotherapy Therapy Dose Expansion-2 (Experimental): - In C-2 (Monotherapy - Advanced or Metastatic Solid Tumors excluding Primary CNS Tumor with or without Brain Metastasis), continuous twice daily oral doses of ABM-1310 at the recommended phase 2 dose (RP2D) from Part A until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion is met.
  Interventions: Drug: ABM-1310
- Combination Therapy Dose Expansion-1 (Experimental): - In C-3 (Combination therapy - Advanced/Metastatic Solid Tumors including Primary CNS tumors but excluding Melanoma with Brain metastasis), continuous twice daily oral doses of ABM-1310 at the recommended phase 2 dose (RP2D) from Part B, in combination with cobimetinib (Cotellic®) 60 mg administered the first 21 days of each 28-day treatment cycle until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion is met.
  Interventions: Drug: ABM-1310; Drug: Cobimetinib
- Combination Therapy Dose Expansion-2 (Experimental): - In C-4 (Combination therapy - Melanoma with Brain Metastasis), continuous twice daily oral doses of ABM-1310 at the recommended phase 2 dose (RP2D) from Part B, in combination with cobimetinib (Cotellic®) 60 mg administered the first 21 days of each 28-day treatment cycle until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion is met.
  Interventions: Drug: ABM-1310; Drug: Cobimetinib

INTERVENTIONS:
Drug: ABM-1310 — Part A: Starting dose at 25 mg by mouth twice daily.
  Part B: Starting dose at a dose below the MTD( Maximum Tolerated Dose) that has been demonstrated to be safe in Part A.
  Part C-1 and C-2: Continuous twice daily oral doses of ABM-1310 at the recommended phase 2 dose (RP2D) from Part A until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion is met.
  Part C-3 and C-4: Continuous twice daily oral doses of ABM-1310 at the recommended phase 2 dose (RP2D) from Part B until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion is met.
  Other Names: ABM1310
Drug: Cobimetinib — Part B: orally administered once daily.
  Part C-3 and C-4: Continuous once daily oral dose from Part B, administered the first 21 days of each 28-day treatment cycle until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion is met.
  Dose formulation is 60 mg capsules.
  Other Names: Cotellic®
  Arms: Combination Therapy Dose Escalation; Combination Therapy Dose Expansion-1; Combination Therapy Dose Expansion-2

SUMMARY:
This is a Phase I, First-In-Human, open label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-cancer activity of ABM-1310 in adult patients with locally advanced or metastatic solid tumors who have no effective standard treatment options available, as monotherapy in patients with documented BRAF V600 mutation, or in combination with cobimetinib (Cotellic®) in adult patients who have documented BRAF mutation and progressive disease or intolerance to at least one prior line of systemic therapy.

DETAILED DESCRIPTION:
This is a Phase I, First-In-Human, open label, dose escalation and dose expansion study to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-cancer activity of ABM-1310 in adult patients with locally advanced or metastatic solid tumors who have no effective standard treatment options available, as monotherapy in patients with documented BRAF V600 mutation, or in combination with cobimetinib (Cotellic®) in adult patients who have documented BRAF mutation and progressive disease or intolerance to at least one prior line of systemic therapy. The primary objectives of this study are to determine the Maximum Tolerated Dose (MTD) and/or the Recommended Phase II Dose (RP2D) of both single agent and combination treatment and to assess the safety and tolerability of ABM-1310 as a monotherapy and in combination.

Study consists of three Parts:

Part A: The starting dose of ABM-1310 is 25 mg po bid, and dose escalation will be guided by a "3+3" design. ABM-1310 will be administered twice daily on a continuous schedule. Each treatment cycle consists of 28 days.

Part B: The starting dose of ABM-1310 will be a dose below the MTD that has been demonstrated to be safe in Part A Monotherapy. A classic "3+3" design will guide the dose escalation. At each dose level, ABM-1310 will be administered in combination with 60 mg cobimetinib (Cotellic ®) once daily (qd) for the first 21 days of each 28-day treatment cycle.

Part C:

* In C-1 (Monotherapy - Primary CNS Tumors) and C-2 (Monotherapy - Advanced or Metastatic solid tumors excluding Primary CNS tumors with or without Brain Metastasis), continuous twice daily oral doses of ABM-1310 at the recommended phase 2 dose (RP2D) from Part A until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion is met.
* In C-3 (Combination therapy - Advanced/Metastatic Solid Tumors including Primary CNS Tumors but excluding Melanoma with Brain Metastsis) and C-4 (Combination therapy - Melanoma with Brain Metastasis), continuous twice daily oral doses of ABM-1310 at the recommended phase 2 dose (RP2D) from Part B, in combination with cobimetinib (Cotellic®) 60 mg administered the first 21 days of each 28-day treatment cycle until disease progression, unacceptable toxicity, or a clinical observation satisfying another withdrawal criterion is met.

Dose limiting toxicity (DLT) will be evaluated and managed per the pre-defined DLT criteria and rules specified in the protocol. MTD and/or RP2D will be confirmed in a dose confirmation cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 18 years and older who are able to sign informed consent and to comply with the protocol
2. Patients with histologically or cytologically-documented, locally advanced, or metastatic solid tumor malignancy that has either (a) progressed on at least one line of prior standard systemic therapy, (b) for which no standard therapy exists, or (c) standard therapy is not considered appropriate by the patient or treating physician. There is no limit to the number of prior treatment regimens

   * Part A: Patients with advanced or metastatic solid tumors with documentation of positive BRAF V600E mutation, or any other BRAF V600 mutation is required for enrollment
   * Part B: Patients with advanced or metastatic solid tumors with documentation of any BRAF mutation.
   * Part C:

     1. C-1: Patients with primary central nervous system (CNS) tumors and documentation of positive BRAF V600 mutation
     2. C-2: Patients with advanced or metastatic solid tumors and documentation of positive BRAF V600 mutation excluding primary CNS tumor
     3. C-3: Patients with advanced or metastatic solid tumors and documentation of positive BRAF mutation including primary CNS tumors but excluding melanoma with brain metastasis
     4. C-4: Patients with melanoma with brain metastasis and documentation of positive BRAF mutation

   Patients with active or stable brain metastasis that are asymptomatic, or that are symptomatic treated with a total daily dose of no more than 4 mg of dexamethasone (or equivalent) that is stable or tapering for at least 2 weeks prior to first treatment are eligible for enrollment. Patients with neurologic signs and symptoms who are not being treated with steroids are eligible and should have no experience of seizure within 2 weeks prior to first treatment.
3. Must have at least one measurable lesion as defined by RECIST V1.1 criteria for solid tumors or the RANO criteria for primary CNS tumors, such as gliomas.

   * For solid tumor with Brain Metastases:
   * Measurable brain lesions that are 0.5 - 3 cm in longest diameter as defined by the modified RECIST V1.1 criteria are allowed.
   * Brain lesion size > 3 cm is not eligible.
4. ECOG performance status of 0 or 1 or Karnofsky performance status of ≥ 70
5. Adequate organ function confirmed at screening and within 28 days of initiating treatment, as evidenced by:

   * Absolute Neutrophil Count (ANC) ≥ 1.0 x 10^9/L
   * Hemoglobin (Hgb) ≥ 9 g/dl
   * Platelets (Plt) ≥ 100 x 10^9/L
   * AST/ALT ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 5.0 x ULN if liver metastases are present
   * Total bilirubin ≤ 1.5 x ULN, or direct bilirubin <ULN for patients with total bilirubin levels >1.5 ULN
   * Serum creatinine <1.5 x ULN or measured or calculated (per institutional standard) creatinine clearance of > 60 mL/min.
6. Negative pregnancy test within 72 hours before starting study treatment in all pre-menopausal women and women <12 months after the onset of menopause
7. Male and female subjects must agree to take sufficient contraceptive methods to avoid pregnancy before first dose of study treatment, during the study, and for at least 3 months after ceasing study treatment

Exclusion Criteria:

1. Women who are pregnant or breast-feeding
2. Women of child-bearing potential (WOCBP) who does not use adequate birth control
3. Patients with any hematologic malignancy. This includes leukemia, lymphoma, and multiple myeloma
4. Have a second primary malignancy that, in the judgment of the investigator, may affect the interpretation of results
5. Patients with carcinomatous meningitis (leptomeningeal disease (LMD))
6. Patients with history of stroke ≤ 6 months prior to starting study drug
7. Patients who have had an experience of seizure within 14 days prior to first treatment
8. Impaired cardiac function or clinically significant cardiac diseases, including but not limited to any of the following:

   * Left Ventricular Ejection Fraction (LVEF) < 45% as determined by MUGA scan or ECHO
   * Congenital long QT syndrome
   * QTcF ≥ 450 msec (mean) on screening (Triplicate 12-Lead ECG)
   * Unstable angina pectoris ≤ 6 months prior to starting study drug
   * Acute myocardial infarction ≤ 6 months prior to starting study drug
   * Use of pacemaker
9. Patients with

   * Unresolved diarrhea ≥ CTCAE Grade 2, or
   * Impairment of gastrointestinal (GI) function, or
   * GI disease or conditions that may significantly alter the absorption of ABM-1310 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
10. Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., uncontrolled hypertriglyceridemia [triglycerides >500 mg/dL], active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
11. Extensive prior radiotherapy to more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation within 5 years
12. Patients who have received chemotherapy, targeted therapy or immunotherapy ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy, except:

    * ≤ 6 weeks for nitrosourea or mitomycin-C
    * ≤ 5 half-lives or 2 weeks for small molecule inhibitor treatment, whichever is longer
13. Patients who have received wide field radiotherapy ≤ 4 weeks, limited field radiation for palliation ≤ 2 weeks, prior whole-brain radiotherapy (WBRT) ≤ 4 weeks or stereotactic radiosurgery (SRS) ≤ 2 weeks (one week for patients with primary CNS tumor such as GBM or with brain metastasis) prior to starting study drug or patients who have not recovered from side effects of such therapy
14. Patients who have undergone major surgery ≤ 4 weeks in general prior to starting study drug or who have not recovered from side effects of such therapy. However, a minimum of 2 weeks recovery time from major surgery prior to starting study drug is acceptable if in investigator's opinion the patient has recovered from surgery.
15. Patients who are currently receiving treatment with therapeutic doses of warfarin sodium or any other coumarin-derivative anticoagulants
16. Patients who have received systemic corticosteroids ≤ 2 weeks prior to starting study drug or who have not recovered from the side effects of such treatment. Therapeutic doses of corticosteroids up to 4 mg/day of dexamethasone, or equivalent are allowed. Note: Patients that are taking replacement doses of steroids are eligible
17. Patients who are currently receiving treatment with medication that has known risk to prolong the QT interval, and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
18. Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory; patients with well controlled HIV might be enrolled per investigator's discretion)
19. Known history of active infection with Hepatitis B (e.g., HBsAg reactive), or Hepatitis C (e.g., S RNA (qualitative) is detected)
20. History of alcohol or drug abuse ≤ 3 months prior to first dose
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that, in the opinion of the investigator, might confound the results of the trial, interfere with the patient's participation and compliance in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) | End of Cycle 1 (each cycle is 28 days) or up to treatment discontinuation (an average of 6 months)
  Determine Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) as a monotherapy and in combination therapy in Part A and Part B
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to study discontinuation (an average of 1 year)
  Safety and tolerability of ABM-1310 as a monotherapy and in combination therapy at Part A and Part B's Recommended Phase 2 dose (RP2D) in Part C
Number of participants with abnormal laboratory values | Up to study discontinuation (an average of 1 year)
  Safety and tolerability of ABM-1310 as a monotherapy and in combination therapy at Part A and Part B's Recommended Phase 2 Dose (RP2D) in Part C

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to 30 days from treatment discontinuation
  Safety and tolerability of ABM-1310 as a single agent and in combination therapy in Part A and Part B
Number of participants with abnormal laboratory values | Up to 30 days from treatment discontinuation
  Safety and tolerability of ABM-1310 as a single agent and in combination therapy in Part A and Part B
Area under the concentration time curve (AUC) | Up to Day 1 of Cycle 2 (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 as a single agent and in combination therapy
Maximum plasma concentration (Cmax) | Up to Day 1 of Cycle 2 (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 as a single agent and in combination therapy
Steady-state concentration (Css) | Up to Day 1 of Cycle 2 (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 as a single agent and in combination therapy
Time to maximum plasma concentration (Tmax) | Up to Day 1 of Cycle 2 (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 as a single agent and in combination therapy
Half-life (T1/2) | Up to Day 1 of Cycle 2 (each cycle is 28 days)
  Pharmacokinetic (PK) profile of ABM-1310 as a single agent and in combination therapy
Objective Response Rate (ORR) | Up to study discontinuation (an average of 1 year)
  Preliminary efficacy of ABM-1310 as a single agent and in combination therapy
Disease Control Rate (DCR) | Up to study discontinuation (an average of 1 year)
  Preliminary efficacy of ABM-1310 as a single agent and in combination therapy
Duration of Response (DOR) | Up to study discontinuation (an average of 1 year)
  Preliminary efficacy of ABM-1310 as a single agent and in combination therapy
Progression free survival (PFS) | Up to study discontinuation (an average of 1 year)
  Preliminary efficacy of ABM-1310 as a single agent and in combination therapy
Overall Survival (OS) | Up to study discontinuation (an average of 1 year)
  Preliminary efficacy of ABM-1310 as a single agent and in combination therapy
Time to Response (TTR) | Up to study discontinuation (an average of 1 year)
  Preliminary efficacy of ABM-1310 as a single agent and in combination therapy

OTHER OUTCOMES:
Exploratory preliminary efficacy in patients by types of BRAF V600 mutation | Up to study discontinuation (an average of 1 year)
  Preliminary efficacy of ABM-1310 as a single agent and in combination therapy
Identification of major metabolite of ABM-1310 in patients who receive ABM-1310 monotherapy in Part C | Up to study discontinuation (an average of 1 year)
  Tests to identify major metabolite of ABM-1310 by a central lab on the post-dose blood samples from patients who receive ABM-1310 monotherapy in Part C

CONTACTS AND LOCATIONS:
Overall Officials: Sarina A Piha-Paul, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (8):
- United States (8):
  - University of California- San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - University of Miami Hospital Sylvester Comprehensive Cancer Center, Miami, Florida
  - Robert H. Lurie Comprehensive Cancer Center (Northwestern University), Chicago, Illinois
  - Henry Ford Cancer Institute, Detroit, Michigan
  - Columbia University Medical Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - UTHealth Science Center Houston Department of Neurosurgery, Houston, Texas

IPD SHARING:
Plan to Share IPD: No